CLINICAL TRIAL: NCT03789656
Title: An Open Label Exploratory Study to Evaluate the Safety, Pharmacokinetics and Efficacy of CRN00808 in Patients With Acromegaly Treated With Somatostatin Analogue Based Treatment Regimens (ACROBAT Edge)
Brief Title: An Study to Evaluate the Safety and Efficacy of Paltusotine for the Treatment of Acromegaly (ACROBAT Edge)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRN00808-03; 2018-002230-20 (EudraCT Number)
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Acromegaly
Keywords: Acromegaly; ACROBAT; EDGE; Paltusotine
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Paltusotine (Experimental)
  Interventions: Drug: Paltusotine

INTERVENTIONS:
Drug: Paltusotine — Paltusotine, capsules, once daily by mouth
  Other Names: CRN00808

SUMMARY:
An open label exploratory study designed to evaluate the safety, efficacy, and pharmacokinetics of paltusotine (formerly CRN00808) in subjects with acromegaly that are treated with somatostatin analogue (SSA) based treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 to 75 years of age
2. Confirmed diagnosis of acromegaly with either a partial or complete response to protocol defined somatostatin analogue therapy regimens
3. Females must be non-pregnant and non-lactating, and either surgically sterile, post-menopausal, or using effective method(s) of birth control
4. Willing to provide signed informed consent

Exclusion Criteria:

1. Treatment naïve acromegaly subjects
2. Prior treatment with paltusotine
3. Pituitary surgery within 6 months prior to Screening. Subjects receiving radiation therapy may be eligible with some restrictions.
4. History or presence of malignancy except adequately treated basal cell and squamous cell carcinomas of the skin within the past 5 years
5. Use of any investigational drug within the past 30 days or 5 half-lives, whichever is longer
6. Positive test at Screening for HIV, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV-Ab) or has a history of a positive result
7. History of alcohol or substance abuse in the past 12 months
8. Any condition that in the opinion of the investigator would jeopardize the subject's appropriate participation in this study
9. Cardiovascular conditions or medications associated with prolonged QT or those which predispose subjects to heart rhythm abnormalities
10. Subjects with symptomatic cholelithiasis
11. Subjects with clinically significant abnormal findings during the Screening Period, and any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardize the subject's safety or ability to complete the study
12. Subjects taking octreotide LAR at a dose higher than 40 mg, or lanreotide depot at a dose higher than 120 mg, or pasireotide LAR at a dose higher than 60 mg
13. Subjects who usually take octreotide LAR or lanreotide depot less frequently than every 4 weeks (e.g. every 6 weeks or 8 weeks)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (6):
  - UCLA Gonda Diabetes Center, Los Angeles, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - OHSU Northwest Pituitary Center, Portland, Oregon
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
- Brazil (3):
  - CETI - Centro de Estudos em Terapias Inovadoras, Curitiba
  - Hospital Universitário Clementino Fraga Filho (HUCFF/UFRJ) Centro de Pesquisa em Neuroendocrinologia, Rio de Janeiro
  - CPQuali Pesquisa Clinica, São Paulo
- LMU Clinic of University of Munich, Munich, Germany
- Greece (4):
  - General Hospital of Athens "Evangelismos", Athens
  - General Hospital of Athens "Gennimatas", Athens
  - General Hospital of Athens "Laiko", Athens
  - General Hospital of Athens "Ippokratio", Thessaloniki
- Hungary (3):
  - Military Health Center, Division of Endocrinology, Budapest
  - Semmelweis University Faculty of Medicine, Budapest
  - University of Pécs Medical School, Pécs
- Azienda Ospedaliera Universitaria Federico II, Napoli, Italy
- New Zealand (2):
  - Waitemata District Health Board, North Shore Hospital, Takapuna
  - Endocrine, Diabetes and Research Centre, Wellington Hospital, Wellington
- Clinic of Endocrinology Independent Public Health Care Centre University Hospital in Kracow, Krakow, Poland
- National Institute of Endocrinology "C. I. Parhon", Bucharest, Romania
- Clinical Centre Serbia, Clinic for Endocrinology, Diabetes and Metabolic Diseases, Belgrade, Serbia
- University Hospital Bratislava, Bratislava, Slovakia
- United Kingdom (2):
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Leeds Teaching Hospitals NHS Trust, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin S, Bender RH, Krasner A, Marmon T, Monahan M, Nelson L. Development and evaluation of the Acromegaly Symptom Diary. J Patient Rep Outcomes. 2023 Feb 15;7(1):15. doi: 10.1186/s41687-023-00541-7. PMID 36792844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 45 subjects were planned to be enrolled in the study. 47 subjects participated in the study.
Pre-assignment Details: A total of 45 subjects were planned to be enrolled in the study. 47 subjects participated in the study.
Groups:
- Group 1: Partial responders on a stable treatment of octreotide long-acting release (LAR) or lanreotide depot (at least 1 Screening IGF-1 value was > upper limit of normal (ULN), and the V2 value was ≤2.5× ULN)
- Group 2: Partial responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and a dopamine agonist (bromocriptine or cabergoline) (at least 1 Screening IGF-1 value was >ULN, and the V2 value was ≤2.5 × ULN).
- Group 3: Complete responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and a dopamine agonist (bromocriptine or cabergoline) (mean of Screening IGF-1 values were ≤ULN).
- Group 4: Complete responders on a stable dose of pasireotide LAR (mean of Screening IGF-1 values were ≤ULN).
- Group 5: Complete responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and pegvisomant (mean of Screening IGF-1 values were ≤ULN).
Period: Screening Period: up to 6 Weeks
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Started | 25 | 10 | 5 | 4 | 3
Completed | 25 | 10 | 5 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period: up to 13 Weeks
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Started | 25 (Treatment Period started with first dose of study drug (10 mg) at V3, approx. 4 wks after last dose of standard acromegaly treatment. During V6/W4 and V9/W7, the dose was titrated up (blinded), if subject was eligible. Dose increase in 10 mg increments were allowed only at V6/W4 (10 mg to 20 mg), V9/W7 (10 mg to 20 mg, or 20 mg to 30 mg), and V12/W10 (10 mg to 20 mg, 20 mg to 30 mg, or 30 mg to 40 mg). No further up-titration was allowed. Daily dose did not exceed 40 mg.) | 10 (Treatment Period started with first dose of study drug (10 mg) at V3, approx. 4 wks after last dose of standard acromegaly treatment. During V6/W4 and V9/W7, the dose was titrated up (blinded), if subject was eligible. Dose increase in 10 mg increments were allowed only at V6/W4 (10 mg to 20 mg), V9/W7 (10 mg to 20 mg, or 20 mg to 30 mg), and V12/W10 (10 mg to 20 mg, 20 mg to 30 mg, or 30 mg to 40 mg). No further up-titration was allowed. Daily dose did not exceed 40 mg.) | 5 (Treatment Period started with first dose of study drug (10 mg) at V3, approx. 4 wks after last dose of standard acromegaly treatment. During V6/W4 and V9/W7, the dose was titrated up (blinded), if subject was eligible. Dose increase in 10 mg increments were allowed only at V6/W4 (10 mg to 20 mg), V9/W7 (10 mg to 20 mg, or 20 mg to 30 mg), and V12/W10 (10 mg to 20 mg, 20 mg to 30 mg, or 30 mg to 40 mg). No further up-titration was allowed. Daily dose did not exceed 40 mg.) | 4 (Treatment Period started with first dose of study drug (10 mg) at V3, approx. 4 wks after last dose of standard acromegaly treatment. During V6/W4 and V9/W7, the dose was titrated up (blinded), if subject was eligible. Dose increase in 10 mg increments were allowed only at V6/W4 (10 mg to 20 mg), V9/W7 (10 mg to 20 mg, or 20 mg to 30 mg), and V12/W10 (10 mg to 20 mg, 20 mg to 30 mg, or 30 mg to 40 mg). No further up-titration was allowed. Daily dose did not exceed 40 mg.) | 3 (Treatment Period started with first dose of study drug (10 mg) at V3, approx. 4 wks after last dose of standard acromegaly treatment. During V6/W4 and V9/W7, the dose was titrated up (blinded), if subject was eligible. Dose increase in 10 mg increments were allowed only at V6/W4 (10 mg to 20 mg), V9/W7 (10 mg to 20 mg, or 20 mg to 30 mg), and V12/W10 (10 mg to 20 mg, 20 mg to 30 mg, or 30 mg to 40 mg). No further up-titration was allowed. Daily dose did not exceed 40 mg.)
Completed | 23 | 10 | 4 | 3 | 3
Not Completed | 2 | 0 | 1 | 1 | 0
Not completed — Prohibited Medication | 1 | 0 | 0 | 1 | 0
Not completed — COVID-19 Lockdown | 0 | 0 | 1 | 0 | 0
Not completed — Unable to Travel | 1 | 0 | 0 | 0 | 0
Period: Follow-up Period: up to 4 Weeks
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Started | 23 | 10 | 4 | 3 | 3
Completed | 22 | 10 | 4 | 3 | 3
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 47 participants who received CRN00808-03, 42 participants completed the trial, 4 participants withdrew from treatment period, and 1 participant withdrew consent during follow up. No participants withdrew due to adverse events.
Groups:
- Group 1: Efficacy Analysis Set - Primary Analysis Population for all efficacy analyses. Only includes participants from Group 1.
  Eligibility to enter this group was specified as: Partial responders on a stable treatment of octreotide long-acting release (LAR) or lanreotide depot (at least 1 Screening IGF-1 value was greater than upper limit of normal (ULN), and the V2 value was ≤2.5× ULN)
- Group 2: Eligibility to enter this group was specified as: Partial responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and a dopamine agonist (bromocriptine or cabergoline) (at least 1 Screening IGF-1 value was >ULN, and the V2 value was ≤2.5 × ULN)
- Group 3: Eligibility to enter this group was specified as: Complete responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and a dopamine agonist (bromocriptine or cabergoline) (mean of Screening IGF-1 values were ≤ULN)
- Group 4: Eligibility to enter this group was specified as: Complete responders on a stable dose of pasireotide LAR (mean of Screening IGF-1 values were ≤ULN)
- Group 5: Eligibility to enter this group was specified as: Complete responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and pegvisomant (mean of Screening IGF-1 values were
  ≤ULN).
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total
Number analyzed (Participants) | 25 | 10 | 5 | 4 | 3 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 8 | 4 | 3 | 2 | 39
  >=65 years | 3 | 2 | 1 | 1 | 1 | 8
Age, Customized [Median (Full Range); unit: years] — (range)
  years
    Age, y, median (range) | 52.0 [31 to 71] | 52.5 [31 to 70] | 51.0 [43 to 69] | 56.0 [46 to 67] | 38.0 [35 to 66] | 51.0 [31 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 3 | 3 | 3 | 27
  Male | 14 | 3 | 2 | 1 | 0 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 2 | 0 | 1 | 13
  Not Hispanic or Latino | 21 | 4 | 3 | 4 | 2 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 5 | 5 | 4 | 3 | 42
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 0 | 0 | 0 | 2
  Other | 0 | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 0 | 2 | 2 | 8
  Germany | 0 | 1 | 0 | 0 | 0 | 1
  Greece | 5 | 0 | 0 | 1 | 0 | 6
  Hungary | 5 | 1 | 0 | 0 | 0 | 6
  Italy | 0 | 0 | 1 | 0 | 0 | 1
  Poland | 2 | 0 | 0 | 0 | 0 | 2
  Romania | 0 | 0 | 0 | 1 | 1 | 2
  Serbia | 3 | 0 | 0 | 0 | 0 | 3
  Slovakia | 1 | 0 | 0 | 0 | 0 | 1
  United Kingdom | 2 | 0 | 0 | 0 | 0 | 2
  Brazil | 4 | 6 | 3 | 0 | 0 | 13
  New Zealand | 0 | 1 | 1 | 0 | 0 | 2
Height [Median (Inter-Quartile Range); unit: centimeter] — Population: Source missing for one participant, data removed and noted as protocol deviation.
  centimeter
    number analyzed (Participants) | 24 | 10 | 5 | 4 | 3 | 46
    (all) | 173.95 [166.50 to 178.50] | 167.75 [160.00 to 173.00] | 173.00 [164.00 to 176.00] | 169.45 [168.45 to 179.65] | 157.50 [155.50 to 169.00] | 170.25 [165.00 to 176.10]
Weight [Median (Inter-Quartile Range); unit: kilogram(s)] — Population: Source missing for one participant, data removed and noted as protocol deviation.
  kilogram(s)
    number analyzed (Participants) | 24 | 10 | 5 | 4 | 3 | 46
    (all) | 90.95 [76.05 to 103.60] | 84.95 [75.00 to 117.00] | 87.30 [79.70 to 88.20] | 107 [88.75 to 114.35] | 77.50 [59 to 82.40] | 87.15 [75.10 to 104.20]
BMI [Median (Inter-Quartile Range); unit: kilogram(s)/square meter] — Population: Source missing for one participant, data removed and noted as protocol deviation.
  kilogram(s)/square meter
    number analyzed (Participants) | 24 | 10 | 5 | 4 | 3 | 46
    (all) | 29.25 [26.30 to 34.15] | 30.30 [27.90 to 38.10] | 28.50 [28.20 to 30.40] | 34.85 [29.55 to 37.25] | 31.20 [20.70 to 34.10] | 29.95 [26.50 to 34.80]
Ring Size [Median (Inter-Quartile Range); unit: Scores on a Scale] — Finger size is an objective measure of soft tissue over-growth and is assessed using the US Ring Size Scale. Measurements are assessed on an increasing scale of US ring sizes scored from 1-17 (smallest to largest), with an increase in ring size between consecutive visits representing increased peripheral swelling. Ring sizers (Tool jewelry sizing tools) were provided to the sites, and sites were instructed to use the same hand and finger at each visit. Population: Source missing for one participant, data removed and noted as protocol deviation.
  Scores on a Scale
    number analyzed (Participants) | 24 | 10 | 5 | 4 | 3 | 46
    (all) | 12.5 [9.5 to 14.5] | 12.0 [9.0 to 12.0] | 11.0 [10.0 to 12.0] | 12.5 [9.5 to 19.0] | 8.0 [8.0 to 9.0] | 12.0 [9.0 to 13.0]
IGF-1 (x ULN) at Baseline [Median (Inter-Quartile Range); unit: ng/mL x ULN] | 1.335 [1.078 to 1.471] | 1.400 [1.214 to 1.650] | 0.922 [0.864 to 0.928] | 0.659 [0.600 to 0.842] | 0.909 [0.806 to 0.964] | 1.214 [0.965 to 1.466]
Serum Growth Hormone Levels [Median (Inter-Quartile Range); unit: nanogram(s)/milliliter] | 0.6907 [0.4910 to 1.5545] | 1.0490 [0.5118 to 1.6127] | 0.8733 [0.7088 to 1.5585] | 0.1976 [0.1518 to 0.6460] | 2.8763 [0.1403 to 10.2843] | 0.8733 [0.4688 to 1.6127]
IGFBP-3 [Median (Inter-Quartile Range); unit: ng/mL] | 0.803 [0.725 to 0.886] | 0.789 [0.736 to 0.899] | 0.684 [0.668 to 0.693] | 0.716 [0.662 to 0.754] | 0.585 [0.540 to 0.788] | 0.786 [0.687 to 0.882]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Median of Screening Values) in Insulin-like Growth Factor-1 (IGF-1) Level
Description: Change from baseline in IGF-1 level at Week 13/End of Treatment (W13/EoT) in Group 1 subjects Efficacy Analysis Set (EAS).
Time Frame: 13 Weeks
Population: Efficacy Analysis Set includes all subjects in Group 1 who received at least one dose of study drug.
Measure: Median (Inter-Quartile Range); unit: ng/mL x ULN
Groups:
- Group 1: Subjects in Group 1 previously treated with octreotide or lanreotide
Arm/Group | Group 1
Number analyzed (Participants) | 25
ng/mL x ULN | -0.034 [-0.107 to 1.07]
Statistical Analysis 1: Comparison: Group 1; The primary efficacy endpoint was completed with the Efficacy Analysis Set (EAS), which included all treated subjects in Group 1. The median (Interquartile range) for change from baseline in IGF-1xULN to Week 13/EoT and p-value from the Wilcoxon signed rank test were presented. Baseline was defined as the mean of all IGF-1xULN values prior to first dose. Last on treatment assessment was used for EoT if subject discontinued before Week 13; Test type: Other; p = 0.6285, Wilcoxon Signed Rank test

2. Secondary Outcome: Proportion of Subjects With Their Last IGF-1 Measurement ≤ Upper Limit of Normal (ULN)
Description: The secondary endpoint was the proportion of participants who maintained IGF-1 response, defined as the last assessment before the EoT with IGF-1 ≤1.0× ULN meet responder criteria, in Group 3, 4, and 5 subjects only at W13/EoT
Time Frame: 13 Weeks
Population: This endpoint was limited to only subjects in Groups 3, 4 and 5 who started the study with IGF-1 ≤ULN.
Measure: Count of Participants; unit: Participants
Groups:
- Group 3: Eligibility to enter this group was specified as: Partial responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and a dopamine agonist (bromocriptine or cabergoline) (at least 1 Screening IGF-1 value was >ULN, and the V2 value was ≤2.5 × ULN)
- Group 4: Eligibility to enter this group was specified as: Complete responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and a dopamine agonist (bromocriptine or cabergoline) (mean of Screening IGF-1 values were ≤ULN)
- Group 5: Eligibility to enter this group was specified as: Complete responders on a stable dose of pasireotide LAR (mean of Screening IGF-1 values were ≤ULN)
Arm/Group | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 5 | 4 | 3
Participants
  Baseline | 5 | 4 | 3
  W13/EoT (Response) | 2 | 1 | 1
  W13/EoT (No Response) | 3 | 3 | 2
Statistical Analysis 1: Comparison: Group 3 vs Group 4 vs Group 5; Test type: Other; p = 0.3877, exact binomial test assuming the null pr; Null proportion = 0.5

3. Secondary Outcome: Proportion of Subjects With Their Last IGF-1 Measurements ≤1.5×ULN
Description: Proportion of participants with IGF-1 ≤1.5× ULN at W13/EoT.
Time Frame: 13 Weeks
Population: This endpoint was estimated for all the subjects in the Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Partial responders on a stable treatment of octreotide LAR or lanreotide depot (at least one Screening IGF-1 value must be >ULN, and the V2 value must be ≤2.5×ULN)
- Group 2: Partial responders on a stable combination treatment of SSA (i.e., octreotide LAR or lanreotide depot) and a dopamine agonist (bromocriptine or cabergoline) (at least one Screening IGF-1 value must be >ULN, and the V2 value must be ≤2.5×ULN)
- Group 3: Eligibility to enter this group was specified as: Partial responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and a dopamine agonist(bromocriptine or cabergoline) (at least 1 Screening IGF-1 value was>ULN, and the V2 value was≤2.5 × ULN)
- Group 4: Eligibility to enter this group was specified as: Complete responders on a stable combination treatment of SRL (ie, octreotide LAR or lanreotide depot) and a dopamine agonist(bromocriptine or cabergoline) (mean of Screening IGF-1 values were ≤ ULN)
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 25 | 10 | 5 | 4 | 3
Participants
  Baseline (Response) | 19 | 6 | 5 | 4 | 2
  W13/EoT (Response) | 20 | 4 | 4 | 3 | 1
  W13/EoT (No Response) | 5 | 6 | 1 | 1 | 2

4. Primary Outcome: Change From Baseline (Median of Screening Values) in Insulin-like Growth Factor-1 (IGF-1) Level
Description: as for outcome 1
Time Frame: 13 Weeks
Population: Efficacy Analysis Set includes all subjects in Group 1 who received at least one dose of study drug.
Measure: Median (Inter-Quartile Range); unit: ng/mL x ULN
Arm/Group | Group 1
Number analyzed (Participants) | 25
ng/mL x ULN
  Baseline | 1.335 [1.078 to 1.471]
  Week 13 (Visit 14)/ End of Treatment | 1.343 [1.169 to 1.448]

ADVERSE EVENTS:
Time Frame: Participants were monitored until the end of the 4-week follow-up period (up to 17 weeks total).
Description: Some participants received uptitrated dose during the treatment period and are therefore counted in multiple dosing groups.
Groups:
- Dose 5 mg: Adverse event occurred when subject was receiving 5 mg dose paltusotine
- Dose 10 mg: Adverse event occurred when subject was receiving 10 mg dose paltusotine
- Dose 20 mg: Adverse event occurred when subject was receiving 20 mg dose paltusotine
- Dose 30 mg: Adverse event occurred when subject was receiving 30 mg dose paltusotine
- Dose 40 mg: Adverse event occurred when subject was receiving 40 mg dose paltusotine
Arm/Group | Dose 5 mg | Dose 10 mg | Dose 20 mg | Dose 30 mg | Dose 40 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/47 | 0/43 | 0/37 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/47 | 1/43 | 0/37 | 0/32
Other Adverse Events (participants affected / at risk) | 0/2 | 23/47 | 24/43 | 15/37 | 19/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 5 mg (N=2) | Dose 10 mg (N=47) | Dose 20 mg (N=43) | Dose 30 mg (N=37) | Dose 40 mg (N=32)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 5 mg (N=2) | Dose 10 mg (N=47) | Dose 20 mg (N=43) | Dose 30 mg (N=37) | Dose 40 mg (N=32)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 6 (6) | 5 (5) | 4 (4) | 7 (7)
Paresthesia (Nervous system disorders) | 0 (0) | 3 (3) | 5 (5) | 2 (2) | 3 (3)
Fatigue (General disorders) | 0 (0) | 5 (5) | 4 (4) | 3 (3) | 4 (4)
Peripheral swelling (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 3 (3) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that PIs cannot publish until the multi-center publication is first published. If no multi-center publication is published within 18 months of the completion date, the PI may publish their results, provided that the Sponsor is given the opportunity to review the proposed publication in advance.

DOCUMENTS (2):
  • Study Protocol (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT03789656/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03789656/SAP_001.pdf